CLINICAL TRIAL: NCT01474330
Title: A Phase 1, Randomized, Double-blind, Placebo Controlled Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Pomalidomide (CC-4047) Following Multiple Daily Doses in Healthy Male Subjects
Brief Title: A Multiple-ascending-dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Pomalidomide (CC-4047) in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CC-4047-CP-006
Record Dates: First submitted 2011-11-16; First posted 2011-11-18 (Estimated); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Healthy
Keywords: Pomalidomide; safety; tolerability; pharmacokinetics
MeSH Terms: interventions — pomalidomide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 0.5-mg Pomalidomide or placebo (Cohort A) (Experimental): A single 0.5-mg pomalidomide capsule or matching placebo administered once daily for 5 days under fasted conditions
  Interventions: Drug: Pomalidomide; Drug: Placebo
- 1-mg Pomalidomide or placebo (Cohort B) (Experimental): This arm may be initiated pending a safety review of Cohort A. A single 1-mg pomalidomide capsule or matching placebo administered once daily for 5 days under fasted conditions.
  Interventions: Drug: Pomalidomide; Drug: Placebo
- 2-mg Pomalidomide or placebo (Cohort C) (Experimental): This arm may be initiated pending a safety review of Cohort B. A single 2-mg pomalidomide capsule or matching placebo administered once daily for 5 days under fasted conditions.
  Interventions: Drug: Pomalidomide; Drug: Placebo

INTERVENTIONS:
Drug: Pomalidomide — 0.5-mg, 1-mg, or 2-mg capsule administered once daily for 5 days under fasted conditions
  Other Names: CC-4047
Drug: Placebo — Placebo capsule

SUMMARY:
To evaluate the safety, tolerability, and pharmacokinetics of pomalidomide administered orally once a day for 5 days, at daily doses of 0.5 mg, 1 mg, or 2 mg.

ELIGIBILITY:
Inclusion Criteria:

Healthy male subjects of any ethnic origin between ages of 18 and 55 with a body mass index between 19 and 30

Exclusion Criteria:

1. Any condition, including the presence of laboratory abnormalities, or psychiatric illness, that would prevent the subject from signing the Informed Consent Document (ICD), places the subject at unacceptable risk if he were to participate in the study, or confounds the ability to interpret data from the study.
2. Presence of any surgical or medical conditions possibly affecting drug absorption, distribution, metabolism, and excretion, or plans to have elective or medical procedures during the conduct of the trial.
3. Exposure to an investigational drug (new chemical entity) within 30 days prior to the first dose administration or 5 half-lives of that investigational drug, if known (whichever is longer).

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2011-08-01 (Actual); Primary Completion 2011-10-01 (Actual); Study Completion 2011-10-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | 28 days after last dose
  Number of participants with adverse events
area under the plasma concentration-time curve | 72 hours after last dose
  area under the plasma concentration-time curve
time to maximum observed plasma concentration | 72 hours after last dose
  time to maximum observed plasma concentration

SECONDARY OUTCOMES:
maximum observed plasma concentration | 72 hours after last dose
  maximum observed plasma concentration
terminal elimination half-life | 72 hours after last dose
  terminal elimination half-life
apparent total plasma clearance | 72 hours after last dose
  apparent total plasma clearance
apparent total volume of distribution, and accumulation ratio | 72 hours after last dose
  apparent total volume of distribution, and accumulation ratio

CONTACTS AND LOCATIONS:
Overall Officials: Maria Palmisano, Study Director — Celgene
Locations (1):
- PPD Phase I Clinic, Austin, Texas, United States